CLINICAL TRIAL: NCT03215394
Title: Evaluation of Social ABCs With Attention Training Intervention for Toddlers With Autism
Brief Title: Evaluation of Social ABCs With Attention Training Intervention for Toddlers With Suspected Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: IWK Health Centre (Other); Dalhousie University (Other); University of Alberta (Other); University of East London (Other); University of London (Other)
Responsible Party: Principal Investigator, Jessica Brian, Psychologist, Clinician Investigator, Holland Bloorview Kids Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-666
Record Dates: First submitted 2017-04-25; First posted 2017-07-12 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Autism Spectrum Disorder
Keywords: Social ABCs; autism; autism spectrum disorder; Early Intervention; Toddler; Early Identification; Pivotal Response Treatment; ASD; PRT; Control Group; treatment Group; At Risk; Social Communication; Positive Affect; Smiling; Social Orienting; Attentional Control; Attentional Disengagement; Naturalistic Developmental Behaviour Intervention; NDBI
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Communication; Smiling | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enhanced Social ABCs (Experimental): Receive 4-week attention training program, followed by 12-week Social ABCs intervention. The stimuli include four gaze-contingent training tasks that will be presented on a laptop screen using custom MATLAB scripts. Each task will be presented until the infant becomes inattentive, at which point they will go to the next task or take a break. Training stimuli will be presented until toddlers become fidgety or distressed.
  Interventions: Behavioral: Attention Training Program; Behavioral: Social ABCs
- Standard Social ABCs (Sham Comparator): Receive 4-week sham attention program, followed by 12-week Social ABCs intervention. Sham attention condition will use identical hardware, administered by the same research staff for the same frequency and duration as the attention training intervention. Infants are exposed to non-gaze contingent visual stimuli that offer no adaptive difficulty levels (infant appropriate television clips and animations). Sham attention stimuli will be presented until toddlers become fidgety or distressed.
  Interventions: Behavioral: Social ABCs; Behavioral: Sham Attention Training
- Treatment As Usual (Other): A convenience sample of age-equivalent toddlers who meet clinical eligibility criteria but are otherwise unable or unwilling to participate in the interventions, will be used as a Treatment as Usual comparison group. The same assessments will be administered at parallel time points through an existing research study. Receive no attention training program and no Social ABCs.
  Interventions: Other: Treatment As Usual

INTERVENTIONS:
Behavioral: Attention Training Program — The attention training involves 8 visits over 4 weeks with pre/post data collection before and after the training, and a follow-up 6 months later. Pre/post data collection involves the ESCS and a Laboratory Temperament Assessment Battery (LabTAB), and a series of on-screen assessment tasks that measure cognitive control, distraction tolerance, sustained attention, habituation, gap-overlap, disengagement, and attention to static images. Training runs from Wk 2-5 with 2 visits per week and is completed in home with the child sitting on the parents lap in front of a monitor. The parent and child are inside a tent to reduce environmental stimuli. The research trainer is outside the tent running the program from a laptop. The program consists of a battery of 9 gaze-contingent training tasks using custom MATLAB scripts. The animated tasks are designed to engage the child and present as developmentally appropriate games. At each visit 6 of the 9 tasks will run for a total of 4min each(24min).
  Arms: Enhanced Social ABCs
Behavioral: Social ABCs — The 6-month Social ABCs parent-mediated intervention consists of 12 weeks of parent training and a 12 week implementation phase. 15 training (parent coaching) sessions are provided by a Research Trainer. Each session with the trainer includes a review of the program manual, practice of the techniques in the child's home, and a 15 min video of the parent-child dyad practicing the intervention. Week 9 and 11 are phone consultations. After the active training is complete, the parent enters the 12-week implementation phase, which includes practicing the techniques on their own, with no trainer instruction or contact. The trainer re-visits the parent and child at Week 24 to collect three 15 min videos; 2 generalization videos are also taken with an untrained examiner.
  Arms: Enhanced Social ABCs; Standard Social ABCs
Other: Treatment As Usual — The Treatment as Usual group acts as a pre-existing convenience sample, consisting of families currently enrolled in a different approved research study run by the same group of investigators. Children in this group have comparable clinical concerns for ASD, and complete the same standardized measures (ADOS, MSEL, ESCS, AOSI) as the Baseline assessment in this RCT, but will not receive Social ABCs or the Attention Training Program. They are able to access any programs or interventions available to them in the general community. This is tracked on a Services Log form, included as part of that study's protocol. Families in this group will have consented to their child's data being shared across studies in this research group.
  Arms: Treatment As Usual
Behavioral: Sham Attention Training — The sham attention condition will use identical hardware, administered by the same research staff for the same frequency and duration as the attention training program (8 visits over 4 weeks including pre/post data collection). In this condition, infants will be exposed to non-gaze contingent visual stimuli that offer no adaptive difficulty levels (ie. clips of age appropriate television shows). Placebo stimuli will be presented until toddlers become fidgety or distressed.
  Arms: Standard Social ABCs

SUMMARY:
The Social ABCs is an evidence-based, developmentally informed, caregiver-mediated behavioural intervention for toddlers with suspected or confirmed Autism Spectrum Disorder (ASD). It is based on principles of Pivotal Response Treatment (PRT, grounded in Applied Behaviour Analysis), and responsive parenting. The two key targets of this program are functional verbal communication and positive caregiver-child affect sharing. This intervention takes place in the context of play and daily routines, and in all contexts is made to be fun, natural and motivating for the child.

In both a pilot study and a recently completed randomized control trial, toddlers whose caregivers received training in the Social ABCs intervention showed significant gains in early language development (both responsivity and initiations), increased child smiling (mediated by parent smiling), and a trend toward increased social orienting (one important manifestation of social attention).

Despite the social-communication benefits demonstrated through the Social ABCs, the research team is also motivated to foster the attentional abilities of toddlers with emerging ASD in response to compelling evidence that early attentional control abilities may play a central role in the emergence of ASD. Based on this knowledge, the current study targets not only social-communication challenges and affect sharing (as per the existing Social ABCs intervention), but also attentional control in toddlers with suspected or confirmed ASD. Using a structured, computerized attention-training protocol, this RCT evaluates the impact of supplementing the standard Social ABCs intervention with pre-intervention attentional control training.

DETAILED DESCRIPTION:
The Social ABCs intervention was developed to meet the need for evidence-based, feasible, and sustainable interventions for toddlers with emerging ASD. Unlike other more comprehensive programs, the Social ABCs selectively targets only two key developmental areas (i.e., functional spoken language and positive affect). These domains were selected in order to promote developmental progress in areas thought to be central at this developmental stage in ASD. By targeting only two core domains, this program maximizes feasibility and portability (i.e., reduces resource demand) while effecting meaningful change with potential for collateral effects in untargeted, but related, areas.

Bolstered by evidence of acceptability, feasibility, and promise from a pilot study, the Social ABCs was subsequently evaluated in a two-site RCT, demonstrating the efficacy of this caregiver-mediated intervention for toddlers with suspected or confirmed ASD. This study found increases in child vocal responsiveness, vocal initiations, parent smiling, and a trend toward increased social orienting in toddlers with suspected or confirmed ASD. Findings also demonstrated that caregivers attained fidelity relatively quickly, rated the intervention as highly acceptable, reported increased feelings of self-efficacy, and did not report increased stress associated with the burden of learning and providing the intervention.

While the Social ABCs intervention effectively targets social-communication skills and positive caregiver-child affect sharing, the previous RCT demonstrated a promising, but non-significant trend toward increased social attention (orienting), which depends on attentional control; the investigators argue that this is another important developmental domain often impaired in ASD. Improving attentional control may reduce or even prevent expression of ASD-related impairments such as emotion dysregulation and impaired social engagement, due to hypothesized relationships in both typical development and ASD. By targeting early attentional control abilities, this research not only also has the potential to enhance understanding of the fundamental mechanisms that drive behavioural dysregulation in ASD, but also to enhance early development in high-risk toddlers.

Wass and Johnson (2011) have successfully used a brief battery of gaze-contingent computer tasks to enhance cognitive control, sustained attention, and attentional disengagement of typically developing infants. This attention training paradigm has now been adapted for use with toddlers with suspected or confirmed ASD, and its impact will be evaluated as part of this study. Participants will be randomized into one of two groups: Enhanced Social ABCs (Social ABCs plus attention training) or Standard Social ABCs (Social ABCs with placebo). A third group, comprised of a convenience sample of age-equivalent toddlers who meet clinical eligibility criteria but are otherwise unable or unwilling to participate in the interventions, will be used as a Treatment as Usual comparison group.

Toddlers in the Enhanced Social ABCs group will receive eight attention training sessions, taking place in-home or in-clinic, which will be twice weekly for four weeks prior to beginning the Social ABCs. The attention training sessions use a computer-based program that is designed to provide practice in disengaging and shifting attention between competing visual stimuli. The Standard Social ABCs group will be allocated to an adjunct sham computer attention training condition in which they will interact with study staff and be exposed to identical computer equipment for the same schedule and duration of visits. However, this paradigm will involve a display of interesting moving on-screen objects without a gaze-contingent component (i.e., placebo). Both programs track the toddlers' gaze behaviours. Toddlers in both conditions will complete the same pre- and post-training testing assessments. The caregivers will be blind to whether children received the attention training or placebo.

Following the attention/placebo phase, caregivers of both groups will receive Social ABCs caregiver coaching with a Social ABCs coach blind to the participants' attention training (vs. placebo) condition. Social ABCs intervention will include 12 weeks of 1.5-hour home visits of tapering frequency, with follow-up visits at key time points. Home visits include a didactic session based on the Social ABCs manual, followed by practice and live coaching (see Brian et al., 2016, for further information).

In response to the 2020 global COVID-19 pandemic, the intervention has shifted to an online format, with sessions being completed virtually with participant families. The delivery schedule and session design remains the same. Follow-up assessment protocol measures that can be collected via mail or virtually are completed at the original time points.

Data from the Treatment as Usual group will be used to compare Standard and/or Enhanced Social ABCs to developmental trajectories of those not receiving this active intervention. These data include scores from standardized measures and eye-tracking data from one portion of the pre- and post-attention training assessments (i.e., a gap-overlap task).

This project is highly relevant to improving early treatment models, and thus, outcomes for toddlers with emerging ASD. Early action capitalizes on brain plasticity, potentially interrupting the negative developmental cascade, and optimizing outcomes in this high-risk group.

ELIGIBILITY:
Inclusion Criteria:

* The child must be 12-30 months of age with clinically significant signs of ASD (must be under 30 months at study enrollment to be included)
* The toddler and parents must live together, and no more than 50km from the study site
* Child is at home with the caregiver at least 50% of the time (no more than 2.5 days a week in child care, nanny, family care, etc.)
* The child must not be involved in other behavioural interventions, such as ABA/IBI and the Hanen programs, for the duration of the study
* The child may participate in no more than 1 hour per week (monthly average) of the following interventions: speech/language, occupational, and physical therapy, for the duration of the study
* The child's diet and medications have not recently been drastically altered, and are not intended to be altered throughout the study.
* The child does not have other neurological disorders (including epilepsy), genetic syndromes that have known association with ASD (e.g., Fragile X syndrome), significant uncorrected sensory impairments (vision, hearing, etc.), or low birth weight (under 2500g).
* The child is not actively experiencing a regression of skills
* The caregiver is conversant in English and could be coached in English
* The child's eyes are successfully tracked with the eye-tracking technology used throughout the study.

Exclusion Criteria:

* Participant fails to meet any of the above listed Inclusion Criteria.

Ages: 12 Months to 30 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Improved Attentional Flexibility | Week 1 (baseline) and Week 6
  Reaction time in Gap-Overlap task (milliseconds)
Improved Attentional Control | Week 1 (baseline) and Week 6
  Percentage of correct trials in a computer-based attention task (%)
Increased Social Orienting to Parent | Week 1 (baseline), Week 6, Week 18, and Week 30
  Percentage of intervals in which child is oriented to caregiver (%)
Increased Child Smiling | Week 1 (baseline), Week 6, Week 18, and Week 30
  Percentage of intervals in which caregiver and child are smiling together (%)
Increased Child Responsivity to Parent Prompt | Week 1 (baseline), Week 6, Week 18, and Week 30
  Gains in proportion of appropriate child vocal responses, following a caregiver prompt (reported as percentage).

SECONDARY OUTCOMES:
Parent Fidelity of Implementation | Week 6, Week 18, and Week 30
  Percentage of intervals during which parents demonstrate appropriate use of the Social ABCs techniques (%)
Receptive Language | Week 0 and Week 30
  Standard score on the Mullen Early Learning Scale (SS)
Expressive Language | Week 0 and Week 30
  Standard score on the Mullen Early Learning Scale (SS)
Joint Attention | Week 0 and Week 30
  Frequency of joint attentions bids on the Mini Early Social Communication (#)Scales

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (3):
  - University of Alberta - Autism Research Centre, Edmonton, Alberta
  - IWK Health Centre / Dalhousie University, Halifax, Nova Scotia
  - Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario
- University of East London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Landry SH, Smith KE, Swank PR. Responsive parenting: establishing early foundations for social, communication, and independent problem-solving skills. Dev Psychol. 2006 Jul;42(4):627-42. doi: 10.1037/0012-1649.42.4.627. PMID 16802896
- [Background] Brian JA, Smith IM, Zwaigenbaum L, Roberts W, Bryson SE. The Social ABCs caregiver-mediated intervention for toddlers with autism spectrum disorder: Feasibility, acceptability, and evidence of promise from a multisite study. Autism Res. 2016 Aug;9(8):899-912. doi: 10.1002/aur.1582. Epub 2015 Dec 21. PMID 26688077
- [Background] Zwaigenbaum L, Bryson S, Rogers T, Roberts W, Brian J, Szatmari P. Behavioral manifestations of autism in the first year of life. Int J Dev Neurosci. 2005 Apr-May;23(2-3):143-52. doi: 10.1016/j.ijdevneu.2004.05.001. PMID 15749241
- [Background] Wass S, Porayska-Pomsta K, Johnson MH. Training attentional control in infancy. Curr Biol. 2011 Sep 27;21(18):1543-7. doi: 10.1016/j.cub.2011.08.004. Epub 2011 Sep 1. PMID 21889346